CLINICAL TRIAL: NCT06991296
Title: Concentration of n-3 PUFA Monohydroxylated Derivatives in Adults With Obesity After Supplementation With "SPM Active®".
Brief Title: Concentration of n-3 PUFA Monohydroxylated Derivatives in Adults With Obesity After n-3 PUFA Supplementation.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Metagenics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24-0328
Record Dates: First submitted 2025-05-19; First posted 2025-05-27 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-05

CONDITIONS: Obesity
Keywords: oxylipins; obesity; fish oil; omega 3 fatty acids; inflammation; Body Mass Index; omega 3 fatty acid supplementation
MeSH Terms: conditions — Obesity; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPM Active® Supplementation (Experimental): All participants will take two SPM Active® soft-gel capsules daily (total 2 g/day) for 12 weeks (± 2-4 days). Fasting blood samples will be drawn at baseline and at end-of-treatment to quantify 14-HDHA, 17-HDHA, and 18-HEPE levels. Validated surveys assessing burnout, life satisfaction, and sleep quality will be administered before and after the supplementation period.
  Interventions: Dietary Supplement: SPM Active®

INTERVENTIONS:
Dietary Supplement: SPM Active® — Participants will take two SPM Active® soft-gel capsules orally each day (total 2 g/day of specialized pro-resolving mediators) for 12 weeks (± 2-4 days). Capsules are provided by Metagenics and contain monohydroxylated n-3 PUFA derivatives (14-HDHA, 17-HDHA, 18-HEPE).

SUMMARY:
The goal of this clinical trial is to learn if daily supplementation with SPM Active® can increase omega 3 polyunsaturated fatty acid derivatives and improve well-being in adults with obesity. The main questions it aims to answer are:

Does 2 g/day of SPM Active® for 12 weeks increase plasma levels of 14-hydroxydocosahexaenoic (HDHA), 17-HDHA, and 18-hydroxy eicosapentaenoic acid (HEPE)?

Does 2 g/day of SPM Active® for 12 weeks improve self-reported burnout, life satisfaction, and sleep quality?

Participants will:

Take two SPM Active® soft-gel capsules daily for 12 weeks (±2-4 days).

Provide 12-hour fasting blood samples before and after the intervention.

Complete validated surveys on burnout, life satisfaction, and sleep quality at baseline and study end.

DETAILED DESCRIPTION:
Purpose: This study aims to explore the effects of 'SPM Active®,' an omega-3 polyunsaturated fatty acid (n-3 PUFA) dietary supplement, on male adults with obesity. The supplement specifically targets the increase of monohydroxylated derivatives of n-3 PUFAs, which play a crucial role in reducing chronic, low-grade inflammation. The primary objective of the study is to determine whether administering SPM Active® at 2g/day for a longer duration (3 months) leads to higher levels of the monohydroxylated derivatives (14-HDHA, 17-HDHA, and 18-HEPE) in adults with obesity (BMI between 30 and 40 kg/m^2, n=33). The secondary objective is to evaluate whether administration of SPM Active® improves the following outcomes: a) burnout, b) life satisfaction, and c) sleep quality. These outcomes will be assessed using validated surveys administered before and after the intervention.

Participants: The study will include 33 healthy male and female participants of any ethnicity, aged 45-60 years, with a BMI of 30-40 kg/m^2.

Procedures: The intervention involves the administration of the dietary supplement 'SPM Active®' provided by Metagenics. All participants will take 2 soft gel capsules per day for 12 weeks, with a window of +/- 2-4 days. A 12-hour fasting blood sample will be collected from each participant before and after the intervention by a licensed phlebotomist at the UNC Nutrition Research Institute (NRI) at Kannapolis, NC. Additionally, participants will complete surveys at the start and end of the study.

ELIGIBILITY:
Inclusion Criteria:

* adults, ages 45-60 years
* Body mass index (BMI) between 30 and 40 kg/m^2
* Any race or ethnicity

Exclusion Criteria:

* Age < 45 years or > 60 years
* pregnant or breastfeeding women
* BMI < 30 kg/m^2 or > 40 kg/m^2
* Diagnosed type 1 or type 2 diabetes
* Active autoimmune disease, liver disease, coagulopathy, or hypothyroidism
* Known allergy to fish or shellfish
* Current use of any of the following medications: asthma controller therapies, anticoagulants, estrogen or testosterone, daily aspirin or NSAIDs.
* Inability to give informed consent
* Receiving immunomodulatory or immunosuppressant therapy
* Known active malignancy or undergoing treatment for malignancy
* Use of n-3 PUFA supplements or high consumption of fatty fish (> 2 servings/week) within 3 months prior to enrollment.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Plasma Levels of Monohydroxylated n-3 PUFA Derivatives (14-HDHA, 17-HDHA, 18-HEPE) | Baseline (Day 0) and End of Treatment (Week 12 ± 2-4 days)
  Mean change from baseline in fasting plasma concentrations of 14-HDHA, 17-HDHA, and 18-HEPE, as quantified by liquid chromatography-mass spectrometry.

SECONDARY OUTCOMES:
Change in Burnout Score | Baseline (Day 0) and End of Treatment (Week 12 ± 2-4 days)
  The assessment of this survey is validated in a systematic review titled, "Maslach Burnout Inventory-General Survey: A Systematic Review and Meta-Analysis of Measurement Properties." This survey is measured on a scale form 0-6 where 0 is never experiencing the stated type of burnout and 6 being experiencing burnout every day. It is divided into three subscale measurements on emotional exhaustion, cynicism, and professional efficacy. High levels of burnout are indicated by high scores in emotional exhaustion and cynicism, along with low scores in professional efficacy.
Change in Life Satisfaction Score | Baseline (Day 0) and End of Treatment (Week 12 ± 2-4 days)
  The life satisfaction survey assesses global life satisfaction and its validity review is conducted by William Pavot and Ed Diener in "The satisfaction With Life Scale and the merging construct of life satisfaction." This survey is measured on a scale of 1-7 where 1 is strongly disagree and 7 is strongly agree. A low score indicates low life satisfaction, whereas a high score indicates a high level of life satisfaction.
Change in Sleep Quality Score | Baseline (Day 0) and End of Treatment (Week 12 ± 2-4 days)
  The sleep quality survey is validated by University of Pittsburgh and is detailed in "The Pittsburgh sleep quality index: a new instrument for psychiatric practice and research." The sleep quality survey is converted to scores, where the scores range form 0-3 with a higher score being indicative of more sleep disturbances.

CONTACTS AND LOCATIONS:
Overall Officials: Saame Shaikh, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Nutrition Research Institute, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: They willl be shared beginning 9 to 36 months following publication of study. Anticipated: December 2025 to March 2028.